CLINICAL TRIAL: NCT05484544
Title: Safety and Efficacy of Hs-cTnT Protocols
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Ulf Ekelund, Professor, Region Skane
Other Study IDs: HscTnTProtocols
Record Dates: First submitted 2022-07-31; First posted 2022-08-02 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-09

CONDITIONS: Chest Pain; Diagnosis
MeSH Terms: conditions — Chest Pain; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biobank bloodsamples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: High sensitivity troponin T — Collection of hs-cTnT samples

SUMMARY:
Chest pain is a common presenting complaint among patients in the emergency department (ED). A large portion of patients with chest pain undergo lengthy assessment in the ED or are admitted to rule out acute oronary syndrome (ACS), often with stress testing, creating a substantial health care burden. The new high-sensitivity cardiac troponin assays allow use of shorter time intervals for repeated blood samples and may improve care for chest pain patients. The aim of this cohort is to evaluate high-sentivity troponin based protocols for ruling out and ruling in ACS in the ED.

DETAILED DESCRIPTION:
This is a prospective observational study conducted at Skåne University Hospital (Lund, Sweden). Patients presenting with non-traumatic chest pain and for whom hs-cTnT testing was ordered at presentation will be enrolled between february 2013 to April 2014 after providing written informed consent. Patients with STEMI during index visit and those with severe communication barriers will not be enrolled. Enrolled patients will have a second blood sample for hs-cTnT analyzed 1 h after the first sample. Patients with hemolysis with a hemoglobin concentration >0.1 g/dl, H-index >=100 in either the 0- or

1-h sample will be excluded. Clinical data and 1-h high sensitivity troponin T samples will be collected by research assistants. Further diagnostic testing and treatment will be performed, as in routine care, at the discretion of the responsible physician.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age
* Presented to the ED with non-traumatic chest pain/discomfort
* Hs-cTnT testing was ordered at presentation

Exclusion Criteria:

* STEMI at presentation
* Severe communication barriers
* Hemolysis with a hemoglobin concentration>0.1 g/dl, H-index>=100

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Consecutive ED chest pain patients
Sampling Method: Probability Sample
Enrollment: 1167 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
30-day MACE | 30 days
  MACE within 30 days including the index visit. MACE was defined as an adjudicated diagnosis of AMI, UA, cardiac arrest, cardiogenic shock, ventricular arrhythmia requiring intervention, atrioventricular block requiring intervention, or death of a cardiac or unknown cause

SECONDARY OUTCOMES:
30-day MACE without UA | 30 days
  Defined as an adjudicated diagnosis of AMI, cardiac arrest, cardiogenic shock, ventricular arrhythmia requiring intervention, atrioventricular block requiring intervention, or death of a cardiac or unknown cause

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Ekelund, Professor, Principal Investigator — Lund University

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be made upon reasonable request

REFERENCES:
- [Background] Mokhtari A, Borna C, Gilje P, Tyden P, Lindahl B, Nilsson HJ, Khoshnood A, Bjork J, Ekelund U. A 1-h Combination Algorithm Allows Fast Rule-Out and Rule-In of Major Adverse Cardiac Events. J Am Coll Cardiol. 2016 Apr 5;67(13):1531-1540. doi: 10.1016/j.jacc.2016.01.059. PMID 27150684
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Aldous SJ, Allen BR, Apple FS, Babel H, Christenson RH, Cullen L, Di Carluccio E, Doudesis D, Ekelund U, Giannitsis E, Greenslade J, Inoue K, Jernberg T, Kavsak P, Keller T, Lee KK, Lindahl B, Lorenz T, Mahler SA, Mills NL, Mokhtari A, Parsonage W, Pickering JW, Pemberton CJ, Reich C, Richards AM, Sandoval Y, Than MP, Toprak B, Troughton RW, Worster A, Zeller T, Ziegler A, Blankenberg S; ARTEMIS study group. Personalized diagnosis in suspected myocardial infarction. Clin Res Cardiol. 2023 Sep;112(9):1288-1301. doi: 10.1007/s00392-023-02206-3. Epub 2023 May 2. PMID 37131096